CLINICAL TRIAL: NCT01594905
Title: A Multicenter, Open-label, Prospective Study to Evaluate Antiviral Efficacy and Safety of Entecavir Plus Tenofovir Combination in Subjects With Multi-drug Resistant Chronic Hepatitis B Virus Infection
Brief Title: Entecavir Plus Tenofovir Combination in Subjects With Multi-drug Resistant Chronic Hepatitis B Virus Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Collaborators: Bristol-Myers Squibb (Industry); Seoul St. Mary's Hospital (Other); The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Sang Hoon Ahn, Associate Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-273
Record Dates: First submitted 2012-05-07; First posted 2012-05-09 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Hepatitis B
Keywords: To explore; adequate management; CHB; Multidrug resistance
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Entecavir 1.0mg + Tenofovir 300mg (Experimental): All subjects will orally take investigational drugs once daily for 48 weeks.
  Interventions: Drug: Entecavir + Tenofovir (MDR group)

INTERVENTIONS:
Drug: Entecavir + Tenofovir (MDR group) — Entecavir 1.0mg + Tenofovir 300mg
  Other Names: Entecavir 1.0mg - Braclude; Tenofovir 300mg - Viread

SUMMARY:
Entecavir(ETV) plus Tenofovir Disoproxil Fumarate(TDF) combination will show effective antiviral activity and prevent further development of antiviral resistance in hepatitis B e antigen(HBeAg)-positive or -negative Chronic Hepatitis B(CHB) patients who experienced multidrug resistance

All subjects will orally take investigational drugs once daily for 48 weeks. All subjects will be assessed at baseline, Week 4, 12, 24, 36 and 48. Evaluations at each visit will include vital signs, physical examinations, laboratory tests and HBV DNA levels. They were also questioned about adverse events and concomitant medications. At baseline and every six months thereafter, serum will be assayed for HBV serology. Genotypic analysis will be performed at baseline and 48 weeks.

DETAILED DESCRIPTION:
1. It has been one of unsolved issues and unmet needs in CHB management to develop an optimal combination regimen to manage multidrug resistant HBV characterized by selection of variants with two or more classes A of signature genotypic resistant mutations1-3
2. Currently adding on Adefovir(ADV) has been generally recommended in Lamivudine(LAM)- or Telbivudine(LdT)-resistant patients but little is known about the optimal management of CHB patients who developed multidrug resistance4
3. Recent report has shown that the combination of LAM plus ADV did not suppress HBV DNA effectively in CHB patients with resistance mutations to both drugs. Only 12.2% of these pts achieved virologic response(VR; HBV DNA <60 IU/mL) at 12 months and multivariable analysis showed that LAM+ADV group and the presence of the rtA181V/T mutation were independently associated with a decreased rate of virologic response (HBV DNA <2,000 IU/ml) at 12 months4
4. ETV has been demonstrated to be effective in patients with ADV resistance but not in patients with proven YMDD mutation. In contrast, TDF has been shown to be effective in patients with YMDD mutation but not necessarily in all patients with ADV resistance.1-3
5. Thus theoretically, the combination of the most potent nucleoside analogue and nucleotide analogue with non-overlapping resistance profiles, such as ETV plus TDF, is expected to be a promising salvage treatment for multidrug resistant HBV but clinical evidence is limited
6. Therefore, this study will explore that adequate management of multidrug resistant patients using ETV plus TDF combination may lead to faster and greater viral suppression and prevent further emergence of antiviral resistance

All subjects will orally take investigational drugs once daily for 48 weeks. All subjects will be assessed at baseline, Week 4, 12, 24, 36 and 48. Evaluations at each visit will include vital signs, physical examinations, laboratory tests and HBV DNA levels. They were also questioned about adverse events and concomitant medications. At baseline and every six months thereafter, serum will be assayed for HBV serology. Genotypic analysis will be performed at baseline and 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 20 years of age
2. History of HBsAg positive for more than 6 months
3. Subject who has a history of genotypic resistance to NAs from two different classes A
4. Detectable HBV DNA (≥ 60 IU/mL) while on any rescue treatment regimen for at least 24 weeks
5. HBeAg-positive and -negative
6. Compensated liver disease (Child-Pugh A)
7. Signed written informed consent after being instructed about the objective and procedure of the clinical study

Exclusion Criteria:

1. Subjects with Alanine Aminotransferase(ALT) > 10xUpper Limit of normal(ULN)
2. Co-infected with hepatitis C virus(HCV) or HIV
3. Pregnant or lactating woman
4. Subject who needs long-term administration of drugs including immunosuppressive agents, agents related to high risk in the hepatic/renal toxicity, agents influencing renal excretion
5. History of liver transplantation or planned for liver transplantation
6. Subject who was diagnosed malignant tumor and has been receiving chemotherapy
7. Subject who has hepatocellular carcinoma(HCC) history or who shows potential HCC finding such as suspicious region in the radiologic exam(abdominal US or CT) or serum Alpha Feto Protein(AFP) elevation
8. Renal Insufficiency (CLcr < 50ml/min based on Cockcroft-Gault equation considering weight, ages and serum creatinine)
9. Patient who has a liver disease other than chronic hepatitis B (e.g. hemochromatosis, Wilson's disease, alcoholic liver disease, nonalcoholic fatty liver disease, alpha 1-antitrypsin deficiency etc.)
10. Subject who has a history of hypersensitivity to study drug or its ingredients
11. Subject who is involved in other clinical trial within 60 days prior to study entry
12. Subject who the investigator deems inappropriate to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieve virologic response(HBV DNA < 60 IU/mL, approximately 300 copies/mL) by real-time PCR at Week 48 | at Week 48
  To evaluate the proportion of subjects who achieve virologic response(HBV DNA < 60 IU/mL, approximately 300 copies/mL) by real-time Polymerase chain reaction(PCR) at Week 48 after Entecavir plus Tenofovir combination therapy

SECONDARY OUTCOMES:
Virologic, serologic, biochemical efficacy and safety profile, as measured by the incidence of clinical adverse events and laboratory abnormalities including renal marker | Week 4, 12, 24, 36, and 48
  To evaluate virologic, serologic and biochemical response and safety of Entecavir plus Tenofovir combination therapy for 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, PhD, Principal Investigator — Yonsei University

REFERENCES:
- [Derived] Park JY, Kim CW, Bae SH, Jung KS, Kim HY, Yoon SK, Han KH, Ahn SH. Entecavir plus tenofovir combination therapy in patients with multidrug-resistant chronic hepatitis B: results of a multicentre, prospective study. Liver Int. 2016 Aug;36(8):1108-15. doi: 10.1111/liv.13059. Epub 2016 Feb 7. PMID 26781724